CLINICAL TRIAL: NCT05383144
Title: Quantitative Evaluation of the Performance of a Deformable Registration Algorithm: Single-center Study Aimed at Implementing a New Off-line Adaptive Radiotherapy Technique in the Treatment of Breast Cancer by Tomotherapy
Brief Title: Deformable Image Registration for Breast Adaptive Tomotherapy
Acronym: DIRB-ATOM
Status: Completed | Type: Observational
Sponsor: Institut de cancérologie Strasbourg Europe (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-001
Record Dates: First submitted 2022-04-28; First posted 2022-05-19 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Other: Complete Positioning scans — Entire treatment zone imaging at mi-treatment and at end of treatment

SUMMARY:
The radiotherapy treatment plan (also called dosimetry) used for all treatment sessions is based on the dosimetric scanner. During the sessions, the anatomy of the breast may vary, and these variations may impact the quality of the treatment. Adaptive radiotherapy is a new technique that allows these changes to be taken into account during treatment by automatically rescheduling the treatment for each session. The proposed trial aims to clinically evaluate one of these adaptive radiotherapy tools (PreciseART) based on deformable registration in order to determine if it can be used in daily practice in the treatment of breast cancer by tomotherapy. The trial will also clarify whether factors, such as duration of treatment, impact the quality of this algorithm.

DETAILED DESCRIPTION:
The dosimetric scanner needed to calculate the dose to be delivered to the tissues will be carried out according to the standard practice. The treatment plan will be carried out by the physicist in accordance with the dose constraints and validated by the radiation therapist. Each treatment session is preceded by positioning imaging to ensure high precision in the treated area. During the first session, the acquisition of the positioning scanner will take into account the entire region of the target volume in accordance with the classic treatment protocol. Usually, the positioning scans of the remaining sessions are carried out on a smaller area around the operating bed in order to reduce the acquisition time. However, in the context of this study, mid- and end-of-treatment positioning scans will be acquired over the same exploration range as on the first day. These scanners will make it possible to compare the contouring work carried out manually by the radiotherapist and that obtained by the deformable registration algorithm.

ELIGIBILITY:
Inclusion Criteria:

Female

* With invasive breast carcinoma (or axillary lymphadenopathy whose pathological examination is compatible with the origin of breast cancer but without an identified primary breast tumor)
* Breast surgery (conservative surgery or mastectomy)
* Treated by (neo)adjuvant chemotherapy or hormonotherapy
* eligible to normo-fractionated breast radiotherapy in 25 sessions of 2 Gray or 15 sessions of 2.67 Gray, associated or not to bed irradiation whatever the delivered dose
* eligible to an irradiation of sus-clavicular, inner mammary chain or axillary lymph nodes
* With helicoidal tomotherapy

Exclusion Criteria:

* Absence of indication for breast radiotherapy
* Absence of indication for lymph nodes irradiation
* partial irradiation of breast
* in situ carcinoma
* intranodal isolated tumor cells
* radiotherapy on prosthesis or surgically reconstructed breast
* antecedent of breast irradiation opr homolateral lymh node irradiation
* bilateral breast cancer

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Adult followed in the context of unilateral breast cancer, treated with chemotherapy and/or neoadjuvant hormone therapy, with partial or total mastectomy and then with adjuvant radiotherapy.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2022-06-27 (Actual); Primary Completion 2023-04-04 (Actual); Study Completion 2023-04-04 (Actual)

PRIMARY OUTCOMES:
Differences between dosimetric metrics on deformed and delineated contours. | Before treatment
  Description of the differences between metrics calculated on delineated contours and contours deformed by artificial intelligence
Differences between dosimetric metrics on deformed and delineated contours. | Mid-treatment : after fraction 7 for patients with 15 fractions (theoretically at day 9) or after fraction 12 for patients with 25 fractions (theoretically at day 16)
  Description of the differences between metrics calculated on delineated contours and contours deformed by artificial intelligence

CONTACTS AND LOCATIONS:
Locations (1):
- Institut de cancérologie Strasbourg Europe, Strasbourg, France